CLINICAL TRIAL: NCT04563273
Title: Randomized, Blinded, Placebo-Controlled Phase I Clinical Trial to Evaluate the Safety and Tolerability of BCG Vaccine for Intradermal Injection in 6-65 Year Olds
Brief Title: Clinical Study of BCG Vaccine for Intradermal Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BCG-I-healthy
Record Dates: First submitted 2020-06-19; First posted 2020-09-24 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Tuberculosis
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy people aged 18-45 (Experimental): Healthy people aged 18-45 has 40 subjects,and it is considered as BCG purified protein derivative(BCG-PPD) skin test and Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10（EC） detection result all negative.
  Interventions: Biological: BCG vaccine 1（0.025mg/0.1ml/person）; Biological: BCG vaccine 2 （0.05mg/0.1ml/person）; Biological: BCG vaccine 3（0.075mg/0.1ml/person）; Biological: BCG vaccine 4 （0.075mg/0.1ml/person）; Biological: Placebo of BCG vaccine （0.1ml/person）
- Healthy people aged 46-65 (Experimental): Healthy people aged 46-65 has 40 subjects,and it is considered as BCG purified protein derivative(BCG-PPD) skin test and Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10（EC） detection result all negative.
  Interventions: Biological: BCG vaccine 1（0.025mg/0.1ml/person）; Biological: BCG vaccine 2 （0.05mg/0.1ml/person）; Biological: BCG vaccine 3（0.075mg/0.1ml/person）; Biological: BCG vaccine 4 （0.075mg/0.1ml/person）; Biological: Placebo of BCG vaccine （0.1ml/person）
- Healthy people aged 11-17. (Experimental): Healthy people aged 11-17 40 subjects,and it is considered as BCG purified protein derivative(BCG-PPD) skin test and Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10（EC） detection result all negative.
  Interventions: Biological: BCG vaccine 1（0.025mg/0.1ml/person）; Biological: BCG vaccine 2 （0.05mg/0.1ml/person）; Biological: BCG vaccine 3（0.075mg/0.1ml/person）; Biological: BCG vaccine 4 （0.075mg/0.1ml/person）; Biological: Placebo of BCG vaccine （0.1ml/person）
- Healthy people aged 6-10 (Experimental): Healthy people aged 6-10 has 40 subjects,and it is considered as BCG purified protein derivative(BCG-PPD) skin test and Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10（EC） detection result all negative.
  Interventions: Biological: BCG vaccine 1（0.025mg/0.1ml/person）; Biological: BCG vaccine 2 （0.05mg/0.1ml/person）; Biological: BCG vaccine 3（0.075mg/0.1ml/person）; Biological: BCG vaccine 4 （0.075mg/0.1ml/person）; Biological: Placebo of BCG vaccine （0.1ml/person）

INTERVENTIONS:
Biological: BCG vaccine 1（0.025mg/0.1ml/person） — Intradermal injection of 0.025mg/0.1ml/person dose BCG.
Biological: BCG vaccine 2 （0.05mg/0.1ml/person） — Intradermal injection of 0.05mg/0.1ml/person dose BCG.
Biological: BCG vaccine 3（0.075mg/0.1ml/person） — Intradermal injection of 0.075mg/0.1ml/person dose BCG.
Biological: BCG vaccine 4 （0.075mg/0.1ml/person） — Intradermal injection of 0.075mg/0.1ml/person dose BCG.
Biological: Placebo of BCG vaccine （0.1ml/person） — Intradermal injection of 0.1ml/person dose Placebo.

SUMMARY:
The study used a randomized, dose-escalation, blinded, placebo-controlled trial design.

In this trial, 160 subjects were enrolled. The test vaccines are divided into four dose groups: dose group 1 (0.025mg / 0.1ml / person), dose group 2 (0.05mg / 0.1ml / person), dose group 3 (0.075mg / 0.1ml / person), dose group 4 (0.1mg / 0.1ml / person), each Each dose group was enrolled according to 18-45、 46-65 、6-10、11-17years old .

The 4 doses are in descending order in the order of 18-45, 46-65, 11-17, and 6-10 years old. Each age group in the same dose group was enrolled in 8 experimental BCG subjects and 2 placebo subjects.

Among subjects aged 6-65 years, the dose group 2 study will be carried out after the safety assessment 14 days after the dose group 1 vaccination, and the dose group 3 study will be carried out after completing the safety assessment 14 days after the dose group 2 vaccination. Dose group 3 studies were carried out after safety assessment 14 days after vaccination. Within the same dose group, after completing the safety assessment 14 days after vaccination for the previous age group, vaccination for the next age group is carried out.

DETAILED DESCRIPTION:
The study used a randomized, dose-escalation, blinded, placebo-controlled trial design.

In this trial, 160 subjects were enrolled. The test vaccines are divided into four dose groups: dose group 1 (0.025mg / 0.1ml / person), dose group 2 (0.05mg / 0.1ml / person), dose group 3 (0.075mg / 0.1ml / person), dose group 4 (0.1mg / 0.1ml / person), each Each dose group was enrolled according to 18-45、 46-65 、6-10、11-17years old .

The 4 doses are in descending order in the order of 18-45, 46-65, 11-17, and 6-10 years old. Each age group in the same dose group was enrolled in 8 experimental BCG subjects and 2 placebo subjects.

Among subjects aged 6-65 years, the dose group 2 study will be carried out after the safety assessment 14 days after the dose group 1 vaccination, and the dose group 3 study will be carried out after completing the safety assessment 14 days after the dose group 2 vaccination. Dose group 3 studies were carried out after safety assessment 14 days after vaccination. Within the same dose group, after completing the safety assessment 14 days after vaccination for the previous age group, vaccination for the next age group is carried out.

BCG-PPD and EC skin test were performed during the screening period, and the skin test results were followed up at 48 hours; blood routine, urine routine, blood biochemistry, HIV antibody test, electrocardiogram, chest X-ray examination, physical examination, vital signs (heart rate, blood pressure) And body temperature), female subjects of childbearing age undergo a blood pregnancy test. Those eligible for entry will receive a dose of the trial vaccine or placebo on the same day (day 0); Observe vital signs (heart rate, blood pressure and body temperature), reactions at the inoculation site, and reactions at the non-inoculation site at 30 minutes, 7 days, and 14 days after vaccination; Blood routine, urine routine, blood biochemistry, electrocardiogram examination on the 14th day after vaccination; BCG-PPD and EC skin tests were performed on the 84th and 180th days after inoculation.

If the blood routine, urine routine, blood biochemistry, electrocardiogram examinations after vaccination are abnormal and have clinically meaningful results, a re-test is required. Under special circumstances, the number of re-tests can be appropriately increased until the follow-up outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6-65 years old, able to provide legal identification;
2. The guardian and/or I agree to participate in this trial, and have the ability to understand the research procedures and sign an informed consent form, and are willing and able to comply with the requirements of the research protocol;
3. The female agrees to have no birth plan within 180 days after participating in the research and voluntarily take effective contraceptive measures;
4. There is no contraindication to BCG vaccination (①Known allergy to any component of this vaccine; ②Patients suffering from acute disease, severe chronic disease, acute episode of chronic disease and fever; ③Immune deficiency, immunocompromised or receiving immunosuppression Treatment; ④patients with encephalopathy, uncontrolled epilepsy and other progressive neurological diseases; ⑤pregnant women; ⑥patients with eczema or other skin diseases), no history of tuberculosis;
5. There are no contraindications to the use of BCG-PPD and EC (patients suffering from acute infectious diseases (such as measles, pertussis, influenza, pneumonia, etc.), acute conjunctivitis, acute otitis media, patients with extensive skin diseases and allergic constitution);
6. According to the medical history, physical examination and laboratory index test results, the investigator judges to be healthy (for example: no history of tumor, abnormal laboratory index but no clinical significance);
7. The average diameter of BCG-PPD 48-hour skin test induration is less than 5mm without double circles, blisters, necrosis and lymphangitis. The average diameter of EC 48-hour skin test induration and redness is less than 5mm without blisters, necrosis, and lymphangitis. reaction.

Exclusion Criteria:

1. Any previous history of severe side effects of vaccines or drugs, such as urticaria, dyspnea, angioedema;
2. The interval between inoculation of live attenuated vaccine is less than 28 days, and the interval of other vaccines is less than 14 days;
3. Those who have a history of convulsions, epilepsy, mental illness and/or family history of mental illness;
4. Human immunodeficiency virus (HIV) antibody test results are positive;
5. Have received blood or blood-related products within 3 months before screening;
6. A history of drug abuse upon inquiry;
7. Women who are breastfeeding;
8. Those who have participated in other clinical trials in the past 3 months and used study drugs;
9. 6-17 years old systolic blood pressure ≥120mmHg and/or diastolic blood pressure ≥80 mmHg; 18-65 years old diastolic blood pressure ≥90mmHg and/or systolic blood pressure ≥140mmHg;
10. Those with axillary body temperature ≥37.3℃;
11. Disabled upper limbs;
12. The researcher believes that the subject has any conditions that may affect the evaluation of the research purpose.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events after vaccination | Up to 6 months after the sixth time injection
  Evaluate safety indicators before vaccination, 30 minutes, 7 days, and 14 days after vaccination. Collect all AEs 30 minutes after vaccination, 0-14 days of collected adverse events, 0-30 days of non-collected adverse events, within 6 months SAE, to evaluate the safety and tolerability of BCG vaccine for intradermal injection used in the test in people aged 6 to 65 years old with negative BCG-PPD and EC skin test

SECONDARY OUTCOMES:
Positive conversion rate of BCG-PPD skin test 12 weeks and 6 months after vaccination | Up to 6 months after the sixth time injection
  BCG-PPD skin tests were conducted 12 weeks and 6 months after inoculation of the corresponding test drugs and placebo to evaluate the positive conversion rate of BCG-PPD after BCG vaccination for intradermal injection
Positive conversion rate of EC skin test 12 weeks and 6 months after vaccination | Up to 6 months after the sixth time injection
  EC skin tests were conducted 12 weeks and 6 months after inoculation of the corresponding test drugs and placebo to evaluate the positive conversion rate of EC after BCG vaccination for intradermal injection

CONTACTS AND LOCATIONS:
Overall Officials: Ting Huang, Master, Principal Investigator — Sichuan Provincial Center for Disease Control and Prevention
Locations (1):
- Sichuan Center for Disease Control and Prevention, Chengdu, Sichuan, China

REFERENCES:
- [Background] Tuberculosis Prevention Trial. Trial of BCG vaccines in south India for tuberculosis prevention. 1979. Indian J Med Res. 2013 Mar;137(3):571. No abstract available. PMID 23776969
- [Background] Expanded programme on immunization. Immunization schedules in the WHO European Region, 1995. Wkly Epidemiol Rec. 1995 Aug 4;70(31):221. No abstract available. English, French. PMID 7662525